CLINICAL TRIAL: NCT02704793
Title: Assessing Clinical Effectiveness of Cerebellar Repetitive Transcranial Magnetic Stimulation (rTMS) on Severity of Motor Signs of Essential Tremor
Brief Title: Cerebellar rTMS for Essential Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Olfati, Dr, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 940597
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — salicylhydroxamic acid; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilateral 1 Hz Cerebellar rTMS (Experimental): Patients will be treated with 900 pulses of 1 Hz rTMS on 90% of resting motor threshold (RMT) delivered over each cerebellar hemisphere for 5 consecutive days.
  Interventions: Other: Bilateral 1 Hz Cerebellar rTMS
- Sham (electrical stimulation) (Sham Comparator): Sham treatment will be performed with the same protocol using a small device placed on the TMS coil (not visible to the patients) producing electrical stimulation (less than 3 mili amperes), to simulate the sensation of real TMS.
  Interventions: Other: Sham (electrical stimulation)

INTERVENTIONS:
Other: Bilateral 1 Hz Cerebellar rTMS — 900 pulses of 1 Hz rTMS on 90% of resting motor threshold (RMT) delivered over each cerebellar hemisphere every day for 5 consecutive days.
  Arms: Bilateral 1 Hz Cerebellar rTMS
Other: Sham (electrical stimulation) — 900 pulses of 1 Hz electrical stimulation (less than 3 mili amperes) delivered over each cerebellar hemisphere every day for 5 consecutive days.
  Arms: Sham (electrical stimulation)

SUMMARY:
Essential tremor (ET) is a low-mortality, though truly burdensome and debilitating condition which is known to be the second most common movement disorder of the adult population only after restless legs syndrome. The prevalence of the disorder in all age groups has been estimated to be 0.9%. Repetitive transcranial magnetic stimulation (rTMS) is an almost safe technique which has been used in diagnosis and treatment of many neurologic and psychiatric conditions. Recent studies have shown that cerebellum has a significant role in development of ET and that rTMS could exert therapeutic effects on its motor symptoms. In this study researchers will recruit at least 30 subjects among patients visiting at the Specialty Clinic of Mashhad Medical University according to researchers exclusion and inclusion criteria and after signing a written informed consent, will randomly be assigned to either real or sham rTMS. On the real rTMS arm, patients will be treated with 900 pulses of 1 Hz rTMS on 90% of resting motor threshold (RMT) delivered over each cerebellar hemisphere for 5 consecutive days and sham treatment will be performed with the same protocol using a small device placed on the TMS coil (not visible to the patients) producing electrical stimulation (less than 3 mili amperes), to simulate the sensation of real TMS. Subject's ear will be protected with earplugs during both real and sham stimulations. After 2 months of follow-up, patients will undergo crossover and receive the other treatment as described above. Patients would be assessed using Fahn-Tolosa-Marin scale at the baseline and again on days 5, 12, and 30 after each real or sham treatment session by a blinded researcher. Data will be analysed by another researcher who is also blind.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of essential tremor (ET) based on Movement Disorder Society criteria, involving at least one hand.
* 18 years or above
* cognitively eligible to give informed consent of participation in the trial.

Exclusion Criteria:

* Cardiac pace-maker or other implanted magnetic device or having other contraindications of performing a routine non-contrast MRI
* skin defect at the occipital area preventing placement of a coil
* Currently pregnant or plan for pregnancy in the next 6 months
* History of seizure
* Other comorbid medical conditions capable of producing or enhancing tremor
* advanced cardiac, renal, hepatic or other disabling conditions making patient physical unable to participate in examination and receiving the intervention
* Use of new drugs with potential effect on tremor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
change in score of Fahn-Tolosa-Marin scale | at the baseline and on days 5, 12, and 30 after each real or sham treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shoeibi, MD, Study Director — Mashhad University of Medical Sciences
Locations (1):
- Department of Neurology, Ghaem Hospital, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided
Considering ethical issues the investigators keep patients' data protected, however these data could be provided for further analysis by other investigators upon acceptance of the Mashhad University of Medical Sciences, Research Ethics Board Committee's subject data protection regulations.